CLINICAL TRIAL: NCT02554045
Title: Effects of Daily Tadalafil on Body Composition in Men With Sexual Distress
Brief Title: Daily Tadalafil on Body Fat and Lean Mass
Acronym: TADBODY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Antonio Aversa, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAAA 801
Record Dates: First submitted 2015-09-08; First posted 2015-09-18 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Sexual Dysfunction
MeSH Terms: conditions — Obesity; Sexual Dysfunction, Physiological | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Active Comparator): Patients will take tadalafil 2.5 mg tablet every morning for 8 weeks and then withdraw tadalafil for 8 weeks
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Patients will take placebo tablet every morning for 8 weeks and then withdraw placebo for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Patients will take tadalafil 2.5 mg tablet every morning for 8 weeks and then withdraw tadalafil for 8 weeks
  Other Names: Cialis
  Arms: Tadalafil
Drug: Placebo — Patients will take placebo tablet every morning for 8 weeks and then withdraw placebo for 8 weeks
  Arms: Placebo

SUMMARY:
Data confirming a role for PDE5 in adipocyte biology in vitro have been recently reported. However, a better understanding of the complex role of PDE5 in fat metabolism and whole body homeostasis requires the use of transgenic animal models either lacking or overexpressing PDE5 in adipose tissue. This will clarify the role of PDE5 in adipose expansion and metabolism, and also in glucose homeostasis and vascular function in vivo. Analysis of expression and activity of PDE5 in different sites of human adipose tissue (i.e. visceral vs. subcutaneous), and also in different metabolic conditions (i.e. high-fat diet vs. low calorie intake) could reveal if PDE5 can be considered to be a reliable 'marker' of metabolic dysfunction of the adipocyte. Importantly, chronic treatment with the PDE5 inhibitor sildenafil in a mouse model of diet-induced insulin resistance caused a significant improvement in insulin sensitivity . Also, in humans chronic exposure to tadalafil confirmed an improvement of insulin sensitivity in men with erectile dysfunction. However, the efficacy of long-term treatment with PDE5i awaits demonstration in human metabolic diseases such as obesity and insulin resistance.

The primary purpose of the study is to investigate the effects of tadalafil taken once a day on body composition in men with sexual distress and/or erectile dysfunction.

DETAILED DESCRIPTION:
Study design: open-label, randomized controlled study Study duration: 16 weeks (8 active treatment + 8 follow-up)

At baseline, after 8 and 16 weeks the following evaluations will be assessed: general physical examination and anthropometric parameters i.e., body weight (BW), height, BMI, and waist circumference (WC). Every eight weeks, body composition was calculated by using a whole body dual-energy X-ray absorptiometry (DEXA-HOLOGIC QDR-1000) according to the instructions of the manufacturer and standardized procedures, and the individual Total Fat Mass (FM) variation has been expressed as delta-variation (%) from baseline. Abdominal fat mass (distrectual, described as R1) was calculated by using arbitrary area of the square chosen by tracing of an ideal line joining last inferior ribs and anterior superior iliac spines. Calibration with the manufacturer's spine phantom and quality control analysis were performed daily. Fat Mass was expressed in grams per square centimeter (g/cm2) and result expressed as variation in percentage. Secondary outcomes were variations forom baseline of IIEF-5, total testosterone, estradiol and testosterone /estradiol ratios.

STATISTICAL EVALUATION With a two-sided alpha value of 5% and power of 90%, a sample size of 20 subjects per arm would be able to detect a 2% variation in the percentage of body lean and fat mass from the baseline at upper waist section (for fat mass) and overall body composition (for lean mass). Also, we tested for the differences between treatment groups by using analysis of variance for repeated measures. Statistical analysis was performed by using the computer statistical package SPSS 11.0 (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects greater than 18 years with any BMI who volunteered to enter the study because of the presence of sexual distress and/or mild erectile dysfunction.

Exclusion Criteria:

* Any concomitant treatment during the prior three months, changes in lifestyle, diet or physical exercise attended within the 16 weeks of study duration; patients actively or potentially trying to start a family or requiring fertility treatment; significant hepatic, respiratory, hematological or renal disease; history of drug or alcohol abuse; history or presence of any cancer; any other reason, which the investigator feels, precludes safe inclusion of the patient.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Variation in lean and fat mass (overall and as evaluated by whole body DEXA Hologic-QDR1000 | 8 weeks
  Changes from baseline in the percentage of lean (overall estimation) and fat mass (abdominal area) and vs. control group as evaluated by whole body dual-energy X-ray absorptiometry (DEXA-HOLOGIC QDR-1000).

SECONDARY OUTCOMES:
Sexual domains (IIEF-5 scores) | 8 weeks
  Variation from baseline and vs control group of the IIEF-5 scores
Body Mass Index (BMI) | 8 weeks
  variation of BMI (Kg/m)
Hormonal variations from baseline and vs control group (Testosterone estradiol levels) | 8 weeks
  Plasma Testosterone and estradiol levels as evaluated by Radioimmunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Aversa, MD-PHD, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aversa A, Fittipaldi S, Bimonte VM, Wannenes F, Papa V, Francomano D, Greco EA, Lenzi A, Migliaccio S. Tadalafil modulates aromatase activity and androgen receptor expression in a human osteoblastic cell in vitro model. J Endocrinol Invest. 2016 Feb;39(2):199-205. doi: 10.1007/s40618-015-0344-1. Epub 2015 Jul 2. PMID 26134065
- [Result] Porst H, Brock GB, Kula K, Moncada I, Montorsi F, Basson BR, Kinchen K, Aversa A. Effects of once-daily tadalafil on treatment satisfaction, psychosocial outcomes, spontaneous erections, and measures of endothelial function in men with erectile dysfunction but naive to phosphodiesterase type 5 inhibitors. J Androl. 2012 Nov-Dec;33(6):1305-22. doi: 10.2164/jandrol.111.015289. Epub 2012 Jul 12. PMID 22790642
- [Result] Aversa A, Caprio M, Antelmi A, Armani A, Brama M, Greco EA, Francomano D, Calanchini M, Spera G, Di Luigi L, Rosano GM, Lenzi A, Migliaccio S, Fabbri A. Exposure to phosphodiesterase type 5 inhibitors stimulates aromatase expression in human adipocytes in vitro. J Sex Med. 2011 Mar;8(3):696-704. doi: 10.1111/j.1743-6109.2010.02152.x. Epub 2010 Dec 22. PMID 21176111